CLINICAL TRIAL: NCT03475303
Title: The Effect of Early Versus Traditional Hospital Discharge on Maternal Outcome for Women Undergoing Elective Cesarean Section
Brief Title: Effect of Early Versus Traditional Hospital Discharge on Maternal Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Heba Saad, principle investigator, Ain Shams university, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Early discharge
Record Dates: First submitted 2018-03-09; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: The Effect of Early Versus Traditional Hospital Discharge for Women Undergoing Elective Cesarean Section

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- early hospital discharge (Experimental): women will be discharged early from hospital 12 hours postoperatively after elective cesarean sections.
  Interventions: Behavioral: early hospital discharge

INTERVENTIONS:
Behavioral: early hospital discharge — early hospital discharge at 8-12 hours for women undergone elective cesarean section

SUMMARY:
This study will investigate the effect of early hospital discharge versus traditional one on maternal outcome for women undergoing elective cesarean sections.

aim of the work is to assess rate of maternal hospital revisits after early hospital discharge at 8-12 hours following elective cesarean delivery compared to the current practice of discharge at 24-48 hours postoperatively.

DETAILED DESCRIPTION:
The effect of early versus traditional hospital discharge on maternal outcome for women undergoing elective cesarean section

Randomized clinical trial

Protocol of a thesis for partial fulfillment of master degree in obstetrics and gynecology

Postgraduate Student: Hebatallah Saad Sedky Mohamed Degree: M.B.B.Ch., faculty of medicine- Alexandria university (2013)

Co-DIRECTOR: Prof. Dr. Ahmed Hamdy Nagiub Abdulrahman Academic Position: professor of Obstetrics and Gynecology Department: faculty of medicine- Ain Shams University

Co-DIRECTOR: Dr. Mohamed Esmat Abbas Shawky Academic Position: Lecturer of Obstetrics and Gynecology Department: faculty of medicine- Ain Shams University

What is already known on this subject? What does this study add? The rate of cesarean delivery is increasing, in developing countries, its rate ranges from 13 to 47% of all cases of delivery (Gibbons et al 2010). Current practice is to discharge women from hospital 24-48 hours after cesarean delivery, however in some rural areas there is a common practice of earlier discharge. The effect of earlier discharge on women health is controversial. The present study will investigate the possibility of earlier discharge to reduce the cost of hospitalization and postoperative care, increase the turnover rate of obstetric hospitals and improve maternal outcome.

Many studies were concerned by early discharge of patients as there is evidence for colorectal surgery suggests that enhanced recovery programmes can reduce hospital stays by 0.5-3.5 days compared with conventional care (Fiona Paton et al 2014).

The average hospital stay following Cesarean delivery in most hospitals is 2 to 4 days (Tan et al 2012). Hospitalization allows close monitoring of women and early discovery and management of complication. Early discharge would, therefore, be a disadvantage and may delay identification and treatment of maternal and infant morbidity (National Institute of Health 2011). In contrast, several studies concluded that early discharge after Cesarean delivery is not associated with maternal readmissions (Brown et al 2011) and is associated with more maternal satisfaction and lesser cost (Umbeli et al 2010) and will decrease burden on medical facilities, increase turnover of obstetrics, reduce the cost of postoperative care, reduce rate of hospital acquired complications and Improve maternal neonatal relationship.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 35 years

  * Gestational age between 37-42 weeks
  * BMI less than 30 kg/m2
  * Have normal uncomplicated pregnancy
  * Planned lower uterine segment Cesarean section
  * Planned for primigravida or previous one or two Cesarean sections
  * Planned to have spinal anesthesia
  * Cesarean sections without intra-operative complications
  * Accepting to participate in the study

Exclusion Criteria:

* • Emergency Cesarean section

  * Gestational age less than 37 or more than 42 weeks
  * BMI 30 kg/m2 or more.
  * Multiple pregnancies
  * Polyhydraminos
  * Abnormal placenta
  * Premature rupture of membranes
  * Previous abdominal surgeries or uterine surgeries
  * Not more than previous two Cesarean sections
  * Anemia: Hemoglobin level less than 10 g/dl
  * Cesarean section with intraoperative complications
  * General anesthesia
  * Fibroid uterus
  * RH incompatibility ( as there maybe delay of availability of anti-d immunoglobulins)
  * History of complicated pregnancy or delivery
  * Medical disorders(hypertension, diabetes mellitus, cardiac, pulmonary, renal, hepatic, endocrine and autoimmune disorders).
  * Women refusing participating in the study
  * Women having any contraindications or refusing spinal anesthesia

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 156 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Rate of maternal hospital revisits | one week postoperatively
  the aim is to reduce rate of maternal hospital revisits after discharge from the hospital which will be assessed by questionnaire

SECONDARY OUTCOMES:
Maternal and family satisfaction, | one week postoperatively
  the aim is to get the maximum satisfaction which will be assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hebatallah S Sedky, M.B.B.Ch, Principal Investigator — Ain Shams University
Locations (2):
- Egypt (2):
  - Ainshams maternity hospital, Cairo, EGY 818
  - Ainshams maternity hospital, Cairo, Egy818

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Adanikin AI, Orji EO, Fasubaa OB, Onwudiegwu U, Ijarotimi OA, Olaniyan O. The effect of post-cesarean rectal misoprostol on intestinal motility. Int J Gynaecol Obstet. 2012 Nov;119(2):159-62. doi: 10.1016/j.ijgo.2012.05.033. Epub 2012 Aug 25. PMID 22925817